CLINICAL TRIAL: NCT07033091
Title: Prevalence of Human Papillomavirus (HPV) in a Healthy Population: A Feasibility Study of Oropharyngeal Cancer Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: National Institute for Cancer Research, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 10000
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Oropharynx Cancer
Keywords: Human Papillomavirus; HPV Infection; oropharyngeal cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Papillomavirus Infections | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants over 40 years attending cooperating dental clinics, who agree to the study, complete questionnaire and provide self-sampled gargling sample. These will be tested by CE-IVD-marked HPV diagnostic test. This arm will include approx. 10000 participants.
  Interventions: Diagnostic Test: Self-sampling by gargling kit at dental clinic; Other: Questionnaire; Diagnostic Test: Blood sampling; Diagnostic Test: Self-sampling of the urogenital area
- Arm B (Experimental): Participants over 40 years selected from available databases receive by mail the study information, questionnaire and self-sampling gargling kit. The kits will be sent back to laboratory and will be tested by CE-IVD-marked HPV diagnostic test. This arm will include approx. 10000 participants.
  Interventions: Other: Questionnaire; Diagnostic Test: Self-sampling by gargling kit at home; Diagnostic Test: Blood sampling; Diagnostic Test: Self-sampling of the urogenital area

INTERVENTIONS:
Diagnostic Test: Self-sampling by gargling kit at dental clinic — Participants will perform a self-sampling at the dental clinic using gargling kit
  Arms: Arm A
Other: Questionnaire — Participants will answer questionnaire online/paper at their home or at the dental clinic
Diagnostic Test: Self-sampling by gargling kit at home — Participants will perform a self-sampling at home using gargling kit
  Arms: Arm B
Diagnostic Test: Blood sampling — Venous blood will be collected from study participants with oral hrHPV positivity, in which the presence of circulating hrHPV DNA will be determined.
Diagnostic Test: Self-sampling of the urogenital area — In case of a positive examination in the oropharynx, the tested individuals will be offered a self-collection HPV examination in the urogenital area (cervicovaginal swab in women or external genital swab in men).

SUMMARY:
This study defines the prevalence of oral infection with high-risk human papillomaviruses (hrHPV) in individuals over 40 years of age in the Czech Republic. It also establishes an effective methodology for oropharyngeal carcinoma screening and optimization of screening and testing procedures.

DETAILED DESCRIPTION:
One of the primary objectives of this study is to clarify the prevalence of oral infection with high-risk human papillomaviruses (hrHPV) in individuals over 40 years of age in the Czech Republic. This research will enable a more precise estimation of the population at risk for oropharyngeal carcinoma, which is essential for the development of targeted preventive and diagnostic strategies.

Another key objective is to establish an effective methodology for oropharyngeal carcinoma screening and to optimize the associated testing procedures. To achieve these goals, participants will be recruited into two predefined cohorts. The first cohort will consist of healthy individuals recruited through cooperating dental and outpatient clinics. The second cohort will involve potential participants identified from available databases (e.g., clinical trial databases, commercial databases, health insurance records), who will be invited to participate via mailed self-collection kits for gargle sampling.

For participants testing positive for oral hrHPV, venous blood samples will be collected at regular intervals to assess the presence of circulating hrHPV DNA. If hrHPV is detected in the oropharynx, participants will be offered self-collection HPV testing of the urogenital tract (cervicovaginal swabs for women or external genital swabs for men).

In both cohorts, the study will evaluate the prevalence of oral (and, if applicable, genital) hrHPV infection, articipation rates, and the return rates of valid samples for hrHPV testing. Additionally, the study will monitor hrHPV persistence and plasma hrHPV DNA in individuals who test positive.

We anticipate that the results of this study will contribute to earlier and more effective diagnosis of oropharyngeal cancer, with potential for significant public health impact by reducing the burden of this disease. For individual participants, involvement in the study may provide an opportunity for clinical follow-up in the event of hrHPV positivity, supporting earlier detection of oropharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 40 years or older at the time of enrollment.
* Individuals who are capable of rinsing the oral cavity by gargling independently.
* Signed informed consent for study participation, molecular-genetic testing, and personal data processing.

Exclusion Criteria:

- Previously diagnosed head and neck cancer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Oral prevalence of high-risk HPV | 24 months
  Prevalence of oral infection with high-risk human papillomaviruses (hrHPV) in the Czech Republic in individuals over 40 years of age will be determined. This will enable a more accurate estimation of the population at risk for oropharyngeal cancer.
Establishment of an effective methodology applicable to oropharyngeal cancer screening | 24 months
  Establishment of an effective methodology applicable to oropharyngeal cancer screening and optimization of the testing procedure to clarify the prevalence of oral infection with high-risk HPV.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, Ph.D., Study Director — Faculty of Medicine and Dentistry, Palacky University, Olomouc
Locations (1):
- Klinika zubního lékařství Fakultní nemocnice Olomouc, Olomouc, Czechia